CLINICAL TRIAL: NCT04182282
Title: Online Training & Certification for Competency in Dementia Friendly Hospital Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HealthCare Interactive, Inc. (Industry)
Collaborators: New York University, New York, NY (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AG044019
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Knowledge, Attitudes, Practice; Burnout, Caregiver; Job Satisfaction
Keywords: Alzheimer's Disease; Dementia; Online Training and Certification; Allied Health Workers; Patient Care; Person-Centered Care; Improved Care
MeSH Terms: conditions — Behavior; Caregiver Burden; Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Wait-list RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate (Experimental): Immediate participants receive the intervention (online training and certification exam) during the study.
  Interventions: Behavioral: CARES Dementia-Friendly Hospitals Online Training and Certification Program
- Control (Experimental): Control participants do not receive the intervention (online training and certification exam) during the study. However, they do receive access to the intervention program (at no cost) at the conclusion of the study.
  Interventions: Behavioral: CARES Dementia-Friendly Hospitals Online Training and Certification Program

INTERVENTIONS:
Behavioral: CARES Dementia-Friendly Hospitals Online Training and Certification Program — The CARES Dementia-Friendly Hospitals Online Training program is a 4-course, 16-module, video-based training program for hospital staff members. The CARES Dementia-Friendly Hospitals Online Certification Program is a 100-point certification exam evaluating knowledge from the online training protocol.

SUMMARY:
This research study will evaluate the CARES Dementia-Friendly Hospitals online training and certification program for Allied Health Workers (nursing assistants, dietary aides, housekeeping employees, hospital transporters, lab/x-ray techs, and unit secretaries) who work in a hospital or medical center.

Participants who sign up for this study will complete two 1-hour assessments (on day 1 and day 45). Participants will be randomly assigned into either an "immediate group" (where Participants complete the online training as part of the research study) or a "control group" (where Participants receive access to the online training at the end of the study). The online training and certification will take Participants approximately 6 hours to complete.

To participate, Participants must be an allied health worker working at a hospital or medical center, have access to a computer/tablet/smart phone with Internet access, be comfortable reading and speaking in English, and age 21 or older.

Deadline to begin the study: January 31, 2020

DETAILED DESCRIPTION:
This randomized control trial (RCT) will evaluate the CARES Dementia-Friendly Hospitals online training and certification program. The study will allow up to 400 Allied Health Workers (nursing assistants, dietary aides, housekeeping employees, hospital transporters, lab/x-ray techs, and unit secretaries) to enroll as research participants from a minimum of 12 hospitals in three different states.

RESEARCH STUDY IMMEDIATE AND CONTROL GROUP STUDY REQUIREMENTS

Participants will be randomly assigned into the immediate training group a the control group.

Immediate training group participants will complete a consent form, an intake evaluation, and have one month to complete the training. At day 45, they will complete an a follow-up evaluation (identical to the intake evaluation).

Control group participants will complete a consent form and an intake evaluation. At day 45, they will complete an a follow-up evaluation (identical to the intake evaluation). Once the study is completed, each Control participant will be giving full access to the CARES Dementia-Friendly Hospitals online training program (at no cost).

MEASURES INCLUDED IN THE PRE- AND POST-EVALUATIONS

The pre- and post-evaluations include assessments on knowledge, attitude, sense of competency, burnout, job satisfaction, and job productivity, all measured with reliable and valid published scales.

TIME TO COMPLETE THE STUDY:

The study will take immediate participants approximately 8 hours to complete. The study will take control participants approximately 2 hours to complete (each will be given voluntary access to the 6-hour program at the end of the study, although this is not a study requirement).

POTENTIAL RISKS:

There are no anticipated associated risks to participants if they sign up for this study. This is an educational program focusing on dementia-friendly hospital strategies.

COSTS:

There is no cost to participate in this study.

INCLUSION REQUIREMENTS:

Participants must be an allied health worker currently working in a hospital or medical center to participate in this study.

Participants must have access to a computer/tablet/smart phone with access to the Internet.

Participants must be comfortable reading and speaking in English.

Participants must be age 21 or older.

ENROLLMENT DEADLINE:

January 31, 2020.

THANK YOU:

Thank you for the interest in this research study. Participation is encouraged from urban, suburban, mid-sized, and rural hospital and medical center staff members.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is an allied health worker currently working in a hospital or medical center to participate in this study.
2. Participant has access to a computer/tablet/smart phone with access to the Internet.
3. Participant is comfortable reading and speaking in English.
4. Participant is age 21 or older.

Exclusion Criteria:

1. Participant is not an allied health worker currently working in a hospital or medical center to participate in this study.
2. Participant does not have access to a computer/tablet/smart phone with access to the Internet.
3. Participant is not comfortable reading and speaking in English.
4. Participant is not age 21 or older.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
32-Item Knowledge Gain Pre-Post Exam | through study completion, an average of 45 days.
  Investigator-developed Knowledge Exam
17-Item Sense of Competence In Dementia Care Staff Questionnaire | through study completion, an average of 45 days.
  Schepers, A. K., Orrell, M., Shanahan, N., & Spector, A. (2012). Sense of competence in dementia care staff (SCIDS) scale: development, reliability, and validity. International psychogeriatrics, 24(7), 1153-1162.
19-Item Approaches to Dementia Questionnaire | through study completion, an average of 45 days.
  Lintern, T., & Woods, B. (1996). Approaches to dementia questionnaire. University of Wales, Bangor, UK.
20-Item Job Satisfaction Questionnaire | through study completion, an average of 45 days.
  Weiss, D. J., Dawis, R. V., & England, G. W. (1967). Manual for the Minnesota satisfaction questionnaire. Minnesota studies in vocational rehabilitation.
26-Item Dementia Questionnaire | through study completion, an average of 45 days.
  McKenzie, G. L., Teri, L., Salazar, M. K., Farran, C. J., Beck, C., & Paun, O. (2011). Relationship between system-level characteristics of assisted living facilities and the health and safety of unlicensed staff. AAOHN Journal, 59(4), 173-180.

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Mittelman, DrPH, Principal Investigator — NYU Langone Medical Center, New York, NY; John V Hobday, MA, Principal Investigator — HealthCare Interactive, Inc.
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CARES Dementia-Friendly Hospitals Online Training and Certification Program — http://www.hcinteractive.com/hospitals